CLINICAL TRIAL: NCT04520555
Title: Comparison of Recovery Profiles Between Flexible Laryngeal Mask Airway and Tracheal Intubation in Nasal Bone Fracture
Brief Title: Flexible Laryngeal Mask Airway Versus Tracheal Intubation in Nasal Bone Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Principal investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-OBS-20-081
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Laryngeal Mask Airway
Keywords: Laryngeal mask airway; Intubation; nasal bone fracture; recovery
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laryngeal mask airway group (Experimental): Flexible laryngeal mask airway is inserted for general anesthesia
  Interventions: Device: Laryngeal mask airway
- intubation group (Active Comparator): Endotracheal intubation was performed for general anesthesia
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Laryngeal mask airway — LMA Flexible is a supraglottic airway device, which can be moved out of the surgical field without displacement of the cuff, or loss of seal for the anesthetist
  Other Names: LMA Flexible,Teleflex Co., Westmeath, Ireland
  Arms: Laryngeal mask airway group
Device: Endotracheal tube — Endotracheal tube is a plain tube, which is most commonly used in general anesthesia.
  Other Names: Portex, Smiths Medical International Ltd., South East England, United Kingdom
  Arms: intubation group

SUMMARY:
In surgery under general anesthesia due to nasal bone fracture, laryngeal mask airway or tracheal intubation has been used. However, it has not been investigated that the difference of recovery profiles according to use of laryngeal mask airway or tracheal intubation in nasal bone fracture surgery. The aim of study is to evaluate the efficacy of the laryngeal mask airway regarding recovery profiles and airway complications, compared to tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists classification 1 or 2 who receive general anesthesia due to nasal bone fracture

Exclusion Criteria:

* Patients with high risk of aspiration, patients who anticipated difficult airway

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
cough during extubation | From end of surgery to extubation
  Grade of cough during periextubation periods (0=no cough, 1=single cough, 2=more than one episode of non-sustained cough, 3=sustained and repetitive cough with head lift)

SECONDARY OUTCOMES:
Adequate tidal volume during mechanical ventilation | From insertion of airway device to extubation
  Tidal volume (ml)
Adequate ventilation during mechanical ventilation | From insertion of airway device to extubation
  end-tidal carbon dioxide
Airway pressure during mechanical ventilation | From insertion of airway device to extubation
  peak and mean airway pressure
Changes of heart rate | Before anethetic induction, 1 minute after intubation, the end of surgery, 1 minute after extubation.
  Heart rate
Changes of blood pressure | Before anethetic induction, 1 minute after intubation, the end of surgery, 1 minute after extubation.
  mean blood pressure
Changes of saturation | Before anethetic induction, 1 minute after intubation, the end of surgery, 1 minute after extubation.
  peripheral saturation
Number of Participants with blood contamination at vocal cord and distal trachea | Between the end of surgery and extubation
  Blood contamination was examined using fibrobronchoscope.
Device blood contamination | At airway device removal
  0=no contamination, 1=external contamination of the tube, 2=some soilage of the inner surface of the tube, 3=frank coating of the inner surface of the tube
Number of Participants with airway complications after extubation | From extubation to 5 minutes after extubation
  laryngospasm, hypoventilation (respiratory rate <8/minutes), desaturation (peripheral pulse oximetry saturation <95%)
Time to eye opening and time to extubation | From anesthetic discontinuation to eye opening and extubation
  Time in seconds from anesthetic discontinuation to eye opening at verbal commend and time in seconds from anesthetic discontinuation to extubation
Number of Participants with postoperative airway complications | 30 minutes after surgery and postoperative 1 day
  Sore throat, hoarseness, dysphagia, and nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: JongYeop Kim, M.D.,Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea